CLINICAL TRIAL: NCT06383156
Title: The Use of Lung Ultrasound, Fluoroscopy and Auscultation to Confirm Proper Positioning of Left Sided Double Lumen Tube: A Comparative Study
Brief Title: The Use of Lung US, Fluoroscopy and Auscultation to Confirm Proper Positioning of Left Sided DLT : A Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD157/2023
Record Dates: First submitted 2023-12-23; First posted 2024-04-25 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-12

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure
Keywords: Ultrasound; Clinical auscultation; Fluoroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auscultation (Active Comparator): correct position of LDLT during single lung ventilation will be confirmed by clinical methods.
  Interventions: Device: Double lumen endotracheal tube
- Ultrasound (Active Comparator): correct position of LDLT during single lung ventilation will be confirmed when lung USG revealed correct lung isolation
  Interventions: Device: Double lumen endotracheal tube
- Fluoroscopy (Active Comparator): correct position of LDLT during single lung ventilation will be confirmed when fluoroscopy visualizes the left bronchial cuff and lumen in left main bronchus.
  Interventions: Device: Double lumen endotracheal tube

INTERVENTIONS:
Device: Double lumen endotracheal tube — correct position of LDLT during single lung ventilation

SUMMARY:
The aim of this study is to compare between The Use of Lung ultrasound, Fluoroscopy and Auscultation to Confirm Proper Positioning of Left Sided DLT in elective thoracic surgeries.

DETAILED DESCRIPTION:
A double - blinded randomized controlled trial, After Approval is obtained from research ethics committee of anesthesia and intensive care department, faculty of medicine, Ain Shams University. the study done over18 months. we included patients age between 18 and 60 years old, Physical status according to American Society Anesthesiology 1-3 that will be scheduled for elective thoracic surgery and who required a left-sided double lumen tube (LDLT) during anesthesia after taking written and informed consent. we excluded anticipated difficult intubation, tracheostomy tube, concurrent pneumothorax, pleural effusion, history of pleurodesis, and/or abnormal pulmonary function test (forced expiration volume in one second, total lung capacity, or forced vital capacity < 50% of the predicted values), BMI > 35 kg/m2 , or < 18kg/m2.

a sample size of at least 30 patients per each group of patients undergoing elective thoracic surgery will achieve 100% power, at alpha error 0.05, by using power analysis and sample size software (PASS 15) (Version 15.0.10) for sample size calculation.

Patients will be randomly allocated into 3 groups utilizing computer generated list for allocation and the group assignments will be placed in a closed envelope.

In Group A, the correct position of LDLT during single lung ventilation will be confirmed by clinical methods.

In Group B, the correct position of LDLT during single lung ventilation will be confirmed when lung USG revealed correct lung isolation.

In Group C, the correct position of LDLT during single lung ventilation will be confirmed when fluoroscopy visualizes the left bronchial cuff and lumen in left main bronchus.

In the three groups correct position of LDLT will be confirmed if there is correct lung isolation by fiberoptic bronchoscopy.

On arrival in the operating room, standard monitoring of the patients' electrocardiogram, pulse oximetry, capnography, and non-invasive blood pressure will be allowed. After preoxygenation with 100% oxygen for 5 minutes, Induction of general anesthesia (GA) was performed by propofol 2 mg/kg and fentanyl 2 μg/kg IV. Laryngoscopy will be facilitated by rocuronium 0.5 mg/kg followed by intubation by DLT according to sex and height. General anesthesia will be maintained using isoflurane 1 - 1.5 Vol.% through positive pressure mechanical ventilation and atracurium top-up doses. All the DLT inserted will be left-sided. Following passage of the endobronchial cuff through the vocal cords, the DLT will be rotated 90 degrees counterclockwise and gently advanced for 28 to 30 cm according to the anesthesiologist's decision and with consideration of the patient's height. Following intubation, both the tracheal and bronchial cuffs will be inflated, and the initial depth of insertion will be recorded.

In group A, assessment of the LDLT position using chest auscultation of the upper and lower chest zones on both sides after tracheal cuff will be initially inflated. This will be followed by inflation of the bronchial cuff and repeated auscultation of the same regions, first with the tracheal lumen clamped and finally with the bronchial lumen clamped.

Correct intubation of the DLT will be confirmed by the existence of symmetrical bilateral lung sounds prior to clamping of the tracheal lumen, then by a reduction in the whole sound of the right lung and the appearance of symmetrical upper and lower lung sounds in the left lung following tracheal lumen clamping. This will be followed by a reduction in the whole sound of the left lung and the appearance of symmetrical upper and lower lung sounds in the right lung following bronchial lumen clamping.

In group B, LUS examination will be performed on both sides of the anterior and lateral chest wall on four quadrants bilaterally in the supine position. LUS scanning will be done in eight areas. The chest areas will be divided on each side into two anterior and two lateral areas. Anterior areas will be outlined from the sternum to the anterior axillary line, while the lateral areas will be from the anterior to the posterior axillary line. Each anterior and lateral area will be further divided into upper and lower areas from the clavicle to the second-third intercostal spaces and from the third space to the diaphragm. The correct position of the DLT will be confirmed with a loss of lung sliding sign on the same clamped lumen side and emergence of lung pulse sign.

In group C, The fluoroscopic device is set to pulsing X-ray beam (1 image/second), low dose, and maximum collimation. The patient is placed as close as possible to the image intensifier. These adjustments resulted in a reduction of absorbed doses. When an incorrect position is encountered after the fluoroscopy, the double lumen tube is relocated under fluoroscopic visualization until the tracheal lumen becomes just above the carina, left bronchial cuff and lumen become in left main bronchus.

In three groups final confirmation of the LDLT position will be done by flexible bronchoscope by blinded expert staff.

The correct DLT placement criteria: (1) the tracheal rings are seen anteriorly and the muscular stria posteriorly, (2) the bronchial cuff is seen below the carina and just above the left bronchus, (3) the tip of the tube is positioned just above the secondary carina through the bronchial lumen.

The incorrect DLT placement criteria: (1) absence of the tracheal rings (esophageal or bronchial intubation), (2) too shallow, defined as more than 50 % of the right bronchus opening is obscured by the bronchial cuff, (3) too deep, defined as either the bronchial cuff after inflation was totally unseen or when the tip of the bronchial tube is seen under the secondary carina.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Physical status: ASA 1-3 that were scheduled for elective thoracic surgery and who required a left-sided double lumen tube (LDLT) during anesthesia after taking written and informed Consent.

Exclusion Criteria:

* Anticipated difficult intubation.
* Tracheostomy tube.
* Concurrent pneumothorax.
* Pleural effusion and emphysema.
* History of pleurodesis, and/or abnormal pulmonary function test (forced expiration volume in one second, total lung capacity, or forced vital capacity < 50% of the predicted values).
* Body mass index more than 35

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-18 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
the specificity in confirming the position of the LDLT and matching the observation of flexible bronchoscope | 2 months after data collection
  The findings collected by the three methods will be checked for its specificity by endobronchial bronchoscopy

SECONDARY OUTCOMES:
sensitivity and accuracy in confirming the position of the LDLT. | 2 months after data collection
  the finding collected by three methods will be checked for its sensitivity by fiberoptic bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: ahmed Morsy, master, Principal Investigator — Anesthesia assistant lecturer ain Shams University